CLINICAL TRIAL: NCT03956758
Title: The Reflexive Logics Structuring the Report to HIV Prevention of MSM Practicing ChemSex in the Context of Circulation of the PreP
Brief Title: HIV Prevention During Chemsex
Acronym: Chemsex
Status: Withdrawn | Type: Observational
Why Stopped: Reclassification by Ethics Committee
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0233
Record Dates: First submitted 2019-05-16; First posted 2019-05-21 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Men Having Sex With Other Men
Keywords: MSM; Chemical sex; HIV prevention; HIV pre-exposure prophylaxis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Semi-directed interview — Semi-directed interview on ChemSex practice

SUMMARY:
In 2016, the number of discoveries of HIV seropositivity is estimated at about 6000 in France. Men who have sex with men (MSM) account for 44% of these infections (68% in the Occitanie region). For the past ten years, there have been new practices of sexual drug use among MSM referred to as Chemsex. These practices expose to sexual risks but also to those related to the consumption of drugs making this population more at risk to get infectious contaminations. In the "PREVAGAY study" conducted in Montpellier in 2015, about 30% of MSM included said they had consumed at least one psychoactive product before or during sex during the last 12 months. In addition, this percentage was significantly higher among HIV-positive men (51% versus 24% of HIV-negative men) and 1% (N = 9) had practiced Slam (Sexual Injection). The results of this study also showed that PreP (Prophylaxis Pre-exposure to HIV) was known by 52% of MSM included and 4% (N = 4) had already used it in the last 12 months. Several observations are needed: many ChemSex users do not use the PreP despite the fact that its effectiveness has been proven in many studies.

The social sciences have been studying the HIV epidemic since its emergence. In the era of HIV chronic disease, the sociologist Gabriel Girard wanted to question the pessimistic observation of epidemiological studies in his thesis work. Some contradictory logics explains this epidemiology of HIV which is maintained, particularly in Montpellier despite the arrival of the PreP.

The main objective of our study is to explore the reflexive logic structuring the report to HIV prevention by MSM practicing ChemSex in Montpellier, in the context of the appearance and dissemination of the PreP.

ELIGIBILITY:
Inclusion Criteria:

* Men who have sex with men (MSM)
* living in Montpellier
* using chemsex drugs at least one during sexual intercourse

Exclusion Criteria:

* under 18 years
* seropositive HIV

Ages: 18 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: MSM living in Montpellier with negative HIV status, having at least one sexual intercourse under drug use during the last 12 months
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
report to HIV | 1 day
  report to HIV contamination during Chemsex

CONTACTS AND LOCATIONS:
Overall Officials: Clemence GIRARD, Medical intern, Principal Investigator — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: Undecided
NC